CLINICAL TRIAL: NCT02023359
Title: Observational Study of Everolimus in Combination With Exemestane in Postmenopausal Patients With Hormone Receptor-positive, HER 2-negative Advanced Breast Cancer
Brief Title: Danish Observational Study of Everolimus Plus Exemestane in Hormone Receptor (HR) Positive, Human Epidermal Growth Factor 2 (HER2) - Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Novartis Healthcare A/S (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001JDK02
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Everolimus and exemestane
  Interventions: Drug: Everolimus and exemestane

INTERVENTIONS:
Drug: Everolimus and exemestane

SUMMARY:
An observational study in patients with advanced ER+, HER2 negative breast cancer, who are treated with everolimus and exemestane in combination. The objective of the study is to assess the safety pattern of everolimus in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with HR-positive, HER2-negative advanced breast cancer who are treated with everolimus and exemestane according to the approved Summary of Product Characteristics (SmPC).
* Patients who started treatment after approval of this indication but before the initiation of this study can be retrospectively included, provided that they have systematically been assessed for adverse events.
* The decision to treat the patient with everolimus and exemestane must be independent of the patient's participation in the study.
* The patient must provide signed Informed Consent before any data can be captured.

Exclusion Criteria:

- No formal exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with HR-positive, HER2-negative advanced breast cancer who are treated with everolimus and exemestane according to the approved SmPC will be included in the study.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 2.5 years

SECONDARY OUTCOMES:
Progression free survival | Up to 2.5 years
Overall response rate | Up to 2.5 years
Clinical benefit rate | Up to 2.5 years
Overall survival | Up to 2.5 years
Time on treatment with everolimus | Up to 2.5 years
Reason for stopping treatment with everolimus | Up to 2.5 years

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aalborg Universitetshospital, Clinical Research unit Department of oncology, Klinik Kirurgi-kræft, Hobrovej 18-22, Aalborg
  - Onkologisk Afdelning, SVS Esbjerg, Esbjerg
  - Department of Oncology, Odense University Hospital, Odense